CLINICAL TRIAL: NCT01987726
Title: Decision Impact Analysis of Foundation Medicine's Next Generation Sequencing Test in Advanced Solid Tumor Malignancies
Brief Title: Comprehensive Gene Sequencing in Guiding Treatment Recommendations Patients With Metastatic or Recurrent Solid Tumors
Status: Completed | Type: Observational
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Collaborators: Foundation Medicine (Industry)
Responsible Party: Sponsor
Other Study IDs: OSU-12067; NCI-2013-00872 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2013-11-13; First posted 2013-11-19 (Estimated); Last update posted 2021-10-28 (Actual); Status verified 2021-10

CONDITIONS: Recurrent Breast Cancer; Recurrent Colon Cancer; Recurrent Rectal Cancer; Stage IV Breast Cancer; Stage IVA Colon Cancer; Stage IVA Rectal Cancer; Stage IVB Colon Cancer; Stage IVB Rectal Cancer
Keywords: Solid Tumor Malignancies
MeSH Terms: conditions — Breast Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tissue, blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational (NGS, FMI testing): PART I: Within 10 weeks of beginning a treatment regimen, tumor tissue samples, Blood Collection and CTCs(Circulating tumor cell)from patients are collected for NGS and FMI testing, respectively. Patients remain on current line of therapy until a change in treatment is warranted. The physician's treatment recommendation is documented prior to the release of the FMI results.
  PART II: Physicians are furnished with FMI test results when patients become eligible for a change in therapy and new treatment recommendations are documented. Treatment is dependent on preferences of the physician, patient, and/or results of the FMI test.
  Interventions: Other: cytology specimen collection procedure; Other: laboratory biomarker analysis

INTERVENTIONS:
Other: cytology specimen collection procedure — Undergo collection of CTCs for NGS and FMI testing, respectively.The most recent tumor sample collected from the patient with enough tissue to perform NGS testing will be selected. Tumor from a metastatic or recurrent cancer lesion is preferred but not required. Tumor collection is for standard of care purposes and thus not detailed in this protocol.For each tissue specimen, a representative H&E stained section will be evaluated by a qualified pathologist to confirm the histopathological diagnosis of cancer and to make a quantitative estimate of the proportion of the specimen that is tumor-related cells and the proportion that is non-tumor cells.
  Other Names: cytologic sampling
Other: laboratory biomarker analysis — 2 tubes of 7.5 mL blood samples each will be collected at time tumor tissue is sent to FMI and sent to Cynvenio Biosystems, Inc for CTC isolation and analysis. Patient CTCs will be recovered using Cynvenio CTC flow cell technology (Cynvenio Biosystems, Inc.) and enumerated using a combination of CD45, DAPI and cytokeratin staining.1 DNA will be isolated from CTCs and amplified using Φ-29 whole genome amplification (GE Healthcare). Sequencing to be performed by FoundationOne™ protocol.
  Other Names: Correlative studies; blood samples

SUMMARY:
This pilot clinical trial studies comprehensive gene sequencing in guiding treatment recommendations in patients with metastatic or recurrent solid tumors. Studying samples of blood and tissue from patients with cancer in the laboratory may improve the ability to plan treatment.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the feasibility and logistics associated with a clinical trial utilizing the Foundation Medicine Incorporated (FMI) test in an academic therapeutic setting.

II. To determine the proportion of patients who will receive a cancer-related therapy based on the results provided by the FMI test.

SECONDARY OBJECTIVES:

I. To explore and report estimates of progression free survival (PFS) of the regimen administered after the FMI test results are revealed and the PFS of the most recent regimen administered before the FMI test results were received.

II. To determine the feasibility of performing Next Generation Sequencing (NGS) on metastatic tumor tissue.

III. To determine the feasibility of administering cancer-related drugs that are proposed by the results of NGS that are not Food and Drug Administration (FDA)-approved for a patient's specific cancer diagnosis.

IV. To collect and report the molecular alterations discovered by NGS of advanced breast and colorectal cancer.

V. To determine in an exploratory manner the concordance of the genomic alterations detected by the FMI test in circulating tumor cells (CTCs) to the genomic alterations detected by FMI test in tumor tissues collected from the same patient.

OUTLINE:

PART I: Within 10 weeks of beginning a treatment regimen, tumor tissue samples and CTCs from patients are collected for NGS and FMI testing, respectively. Patients remain on current line of therapy until a change in treatment is warranted. The physician's treatment recommendation is documented prior to the release of the FMI results.

PART II: Physicians are furnished with FMI test results when patients become eligible for a change in therapy and new treatment recommendations are documented. Treatment is dependent on preferences of the physician, patient, and/or results of the FMI test.

After completion of study, patients are followed up for at least 18 months.

ELIGIBILITY:
Inclusion Criteria:

* Are able to understand and provide written informed consent (most recent patient informed consent form) prior to initiation of any study-specific procedures
* Patients are diagnosed with recurrent or metastatic a solid tumor cancer; the first patients to be enrolled will have a diagnosis of breast cancer (Cohort 1) or colorectal cancer (Cohort 2)
* Patients may enter this study at any line of therapy
* Patients must have a tumor sample available for NGS testing
* Patients are within 10 weeks of starting their current line of therapy and enrolled before their 1st computed tomography (CT) scan
* Have an expected survival of >= 3 months, as estimated by the treating oncologist
* Have an Eastern Cooperative Oncology Group performance status (ECOG PS) of 0-2

Exclusion Criteria:

* Are pregnant or nursing women
* Are unable to comply with requirements of the study
* Have a serious uncontrolled intercurrent medical or psychiatric illness, including serious infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with recurrent or metastatic a solid tumor cancer.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2013-09-03 (Actual); Primary Completion 2021-06-10 (Actual); Study Completion 2021-06-28 (Actual)

PRIMARY OUTCOMES:
Feasibility of NGS on metastatic solid tumor tissue, in terms of number of patients screened, FMI test attempted, FMI test successful, and FMI tests results released to physicians | Up to 18 months
  Summary tables will be generated.
Feasibility of NGS result-based non-FDA-approved treatment plan, measured by reasons for ability or inability to receive an anti-cancer agent | Up to 18 months
  Summary tables will be generated.
Availability of recommended experimental regimens via clinical trials | Up to 18 months
Proportion of patients who have one recommended therapy | Up to 18 months
  The proportion of patients who have one recommended therapy recommended will be assessed and compared with the proportion who have multiple options recommended. Summarized, and estimates derived along with corresponding 95% confidence intervals.
Proportion of patients who have multiple options recommended | Up to 18 months
  The proportion of patients who have one recommended therapy recommended will be assessed and compared with the proportion who have multiple options recommended. Summarized, and estimates derived along with corresponding 95% confidence intervals.

SECONDARY OUTCOMES:
Presence of any oncogene or tumor suppressor gene mutations or amplifications identified by NGS on tumor tissue in each cohort | Up to 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Maryam Lustberg, MD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Arthur G. James Cancer Hospital and Solove Research Institute at Ohio State University Medical Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Adams EJ, Asad S, Reinbolt R, Collier KA, Abdel-Rasoul M, Gillespie S, Chen JL, Cherian MA, Noonan AM, Sardesai S, VanDeusen J, Wesolowski R, Williams N, Shapiro CL, Macrae ER, Pilarski R, Toland AE, Senter L, Ramaswamy B, Lee CN, Lustberg MB, Stover DG. Metastatic breast cancer patient perceptions of somatic tumor genomic testing. BMC Cancer. 2020 May 6;20(1):389. doi: 10.1186/s12885-020-06905-2. PMID 32375690
- See also: The Jamesline — http://cancer.osu.edu